CLINICAL TRIAL: NCT00722462
Title: The Effect of Acupuncture on Pregnancy Rates in Women Undergoing Embryo Transfer After in Vitro Fertilization: A Prospective Randomized Sham-controlled Trial
Brief Title: The Effect of Acupuncture on Pregnancy Rates in Women Undergoing Embryo Transfer
Acronym: AcuIVF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recent abstract publication questioning the need for our study
Sponsor: Ottawa Fertility Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OttawaFC
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Pregnancy
Keywords: Infertility; IVF; Acupuncture
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Active acupuncture
  Interventions: Procedure: Active acupuncture
- 2 (Sham Comparator): Sham Acupuncture- acupuncture at neutral points
  Interventions: Procedure: Sham acupuncture
- 3 (No Intervention): Embryo transfer with no acupuncture

INTERVENTIONS:
Procedure: Active acupuncture — Acupuncture 25 minutes before and after embryo transfer
  Arms: 1
Procedure: Sham acupuncture — Acupuncture at neutral points, 25 minutes before and after embryo transfer
  Arms: 2

SUMMARY:
The present study is designed to test the hypothesis that acupuncture, before and after embryo transfer, significantly improves pregnancy rates, compared to embryo transfer with sham acupuncture and no acupuncture at all.

ELIGIBILITY:
Inclusion Criteria:

* patient is undergoing embryo transfer after IVF or ICSI
* patient has given informed consent to participate

Exclusion Criteria:

* frozen embryo transfer
* previous enrollment in study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy | 4-5 weeks after treatment

SECONDARY OUTCOMES:
Live birth | 9 months after treatment
Implantation rate | 4-5 weeks after treatment
Side effects with acupuncture treatment | 2 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Leader, MD, Study Chair — Ottawa Fertility Centre; Doron Shmorgun, MD, Principal Investigator — Ottawa Fertility Centre
Locations (1):
- Ottawa Fertility Centre, Ottawa, Ontario, Canada